CLINICAL TRIAL: NCT02436772
Title: Utilization of the OncoCEE™ Platform to Evaluate Selected Biomarker Alterations in CTCs Isolated From Patients With MBC
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: SCRI HEOR_05
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the performance of a blood test for detecting biomarkers in metastatic breast cancer patients at one clinic against standard testing.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to detect the expression of FGFR1 and AR on circulating tumor cells (CTCs) isolated from the peripheral blood of metastatic breast cancer (MBC) patients using the OncoCEE™ platform. No procedures will be associated with this study, as these mutations will be evaluated from the leftover blood that has already been sent for standard of care ER and HER2 using the same platform. Results from this testing will be correlated with results obtained from standard testing to calculate the rate of concordance between tests.

ELIGIBILITY:
Inclusion Criteria:

* Current patient at participating clinic
* Metastatic breast cancer diagnosis
* 18 years of age or older

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 metastatic breast cancer patients from 1 clinic in Tennessee
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Concordance with standard test | 6 months
  determined by the comparison between OncoCEE test and conventional test

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hamilton, MD, Principal Investigator — SCRI
Locations (1):
- Tennessee Oncology, Nashville, Tennessee, United States